CLINICAL TRIAL: NCT04411563
Title: The Effect of miRNA and Epigenetic Modifications on Prognosis in Covid-19 Infection
Brief Title: Epigenetic Tools as Prognostic Predictors in Covid19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Gokhan Tolga Adas, Faculty Member, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2020/143
Record Dates: First submitted 2020-05-25; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Prognosis
Keywords: COVID 19; Prognostic Epigenetics; miRNA; DNA methylation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Biospecimen Retention: Samples With DNA — Genomic material will be stored to continue prognostic biomarker studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I-Mild: The patients who have these mild symptoms are low-grade fever (not more than 38 degrees celsius), dry cough, fatigue, sore throat, headache, the new loss of taste, and smell. Patients with normal or mild pneumonia findings of radiological imaging and blood lymphocyte count ≥800 / µl and serum CRP≤40 mg /l, ferritin ≤500ng/ml, D-Dimer ≤1000 ng/ml will be included in group I.
  Interventions: Other: Taking biological samples
- Group II-Moderate: The patients who have these moderate symptoms are fever of about 38,5-39 degrees celsius, chills, deep cough, fatigue and body aches, muscle pain, the general feeling of being unwell. Patients with bilateral diffuse pneumonia findings of radiological imaging or blood lymphocyte count <800 / µl or serum CRP> 40 mg / l or ferritin> 500ng / ml or D-Dimer> 1000 ng / ml will be included in group II.
  Interventions: Other: Taking biological samples
- Group III-Severe: The patients who have these severe symptoms are all the common symptoms mentioned above along with shortness of breath, chest discomfort, confusion/unresponsiveness, bluish face/lips, possible gastrointestinal issues, like diarrhea or nausea. Patients with ICU (intensive care unit) admission criteria, such as confusion or tachycardia (> 125 / min) or respiratory distress or tachypnea (> 22 / min) or hypotension <90/60 mmHg or SPO2 <93%will be included in group III. Also, patients with the central nervous system and heart involvement will be directly included in the severe case group
  Interventions: Other: Taking biological samples

INTERVENTIONS:
Other: Taking biological samples — Taking blood samples for biochemical and epigenetic analysis

SUMMARY:
The necessity for early detection and hence improving the outcome of treatment of pneumonia is critical especially SARS-CoV-2 induced cases. This work was designed to evaluate the potential application of measuring circulating epigenetic markers namely, miR-744, miR-24, miR-124, miR-155, miR-19a, miR-122, miR-21, miR-223, let-7f, miR-146, miR-196, miR-136, P13-K, miR-9 expression, and DNA methylation profiling of the ACE2, TMPRSS2, PARP, HOX1 genes in Coronavirus disease 2019 (COVID-19) due to SARS-CoV-2 with/without pneumonia and severe acute respiratory syndrome (SARS) patients as an attempt to evaluate the potential benefits of these new circulating, prognostic, epigenetic markers for Turkish patients.

DETAILED DESCRIPTION:
The objectives of this observational study are 1) To investigate why COVID-19 infection causes different biological behavioral patterns in individuals, 2) To determine the role of epigenetic mechanisms here to detect the difference between individuals, 3)To determine the effectiveness of this behavior model and mechanisms on clinical treatment and to ensure that the results obtained are a step for further treatment studies, 4) To evaluate whether the data obtained in MicroRNA analysis is a predictive marker on prognosis. Material and methods Study design This is an observational prospective cohort study. In the power analysis performed with the G * power 3.1 programs related to our study, the effect size for the lymphocyte percentage and C-reactive protein was found to be 0.57 (Effective Treatment of Severe COVID-19 Patients with Tocilizumab) (alpha probability of error = 0.05); in the sample width analysis, taking the power value 0.80, the total number of patients to be collected was 105 (105/3 = 35 for each group).

Patient's criteria This study was approved by the Clinical Research Ethics Committee (2011- CREC-40) at Bakırköy Dr.Sadi Konuk Training and Research Hospital and informed consent will be obtained from all patients according to the rules of the Declaration of Helsinki. Approval of the local ethical committee number is 2020/143 (2011-CREC-40). Patients enrolled in this study will be admitted to the Infectious Diseases and Clinical Microbiology Department and the Intensive Care Department from May 2020 to September 2020. Diagnosis of COVID 19 will be depending upon the presence of specific lesions in lungs confirmed by computed tomography (CT), and/or laboratory findings according to the Republic of Turkey Ministry of Health diagnostic criteria.

Inclusion criteria All patients between the ages of 18 and 65 included will suffer from COVID 19, and specific treatment should not yet be initiated. COVID 19 diagnosis of patients will be based on full medical history, thorough clinical examination, radiological imaging, laboratory assessment, and SARS-CoV-2 analysis by RT-PCR.

Exclusion criteria

1. People with chronic lung disease or previous AC surgery
2. People with immune deficiency or cancer patients
3. Patients receiving immunosuppressive therapy for autoimmune disease
4. People with neurological diseases affecting the respiratory muscles, such as hypotonia.

On the basis of the inclusion and exclusion criteria 105 patients subjects will be included in this study, divided into three groups; group I (n = 35) patients are mild, group II (n = 35) patients are moderate, and group III (n = 35) patients are severe and critical. Mild and moderate cases are usually defined as those without severe pneumonia or severe acute respiratory syndrome. Mild symptoms are low-grade fever (not more than 38 degrees celsius), dry cough, fatigue, sore throat, headache, the new loss of taste, and smell. Patients with normal or mild pneumonia findings of radiological imaging and blood lymphocyte count ≥800 / µl and serum CRP≤40 mg /l, ferritin ≤500ng/ml, D-Dimer ≤1000 ng/ml will be included in group I. Moderate symptoms are fever of about 38,5-39 degrees celsius, chills, deep cough, fatigue and body aches, muscle pain, the general feeling of being unwell. Patients with bilateral diffuse pneumonia findings of radiological imaging or blood lymphocyte count <800 / µl or serum CRP> 40 mg / l or ferritin> 500ng / ml or D-Dimer> 1000 ng / ml will be included in group II. Severe symptoms are all the common symptoms mentioned above along with shortness of breath, chest discomfort, confusion/unresponsiveness, bluish face/lips, possible gastrointestinal issues, like diarrhea or nausea. Patients with ICU (intensive care unit) admission criteria, such as confusion or tachycardia (> 125 / min) or respiratory distress or tachypnea (> 22 / min) or hypotension <90/60 mmHg or SPO2 <93%will be included in group III. Also, patients with the central nervous system and heart involvement will be directly included in the severe case group.

Specimen collection and handling About 10 ml of peripheral venous blood will be collected under strict aseptic conditions by clean venipuncture using vacuum blood collection tubes and will be distributed as 3 ml in EDTA tubes for complete blood count and DNA extraction, 3 ml in another sterile special RNA protective tube (stored at -80 °C) for miRNA extraction. In addition, 4 ml in a plane tube will be allowed to clot at the room temperature and then will be centrifuged at 3000 rpm for 10 minutes and the collected serum will be stored at -80°C to be used for analyzing cytokine, and other specific tests.On the 7th day of treatment, second samples will be taken under the same conditions and finally, on the 21st day, third samples will be taken.

Laboratory investigations RNA Extraction was done according to the miRNeasy Serum/Plasma Advanced Kit (cat. no. 217204) https:// www.qiagen.com/

The expressions of selected miRNAs and genes were analyzed using Real-Time PCR. The list of required kits, chemicals and consumables is as follows:

miRCURY LNA RT Kit (Cat No: 339340) miRCURY LNA miRNA PCR Assay (200) (Cat No: 339306) miRCURY LNA SYBR Green PCR Kit (600) (Cat No: 339346) miRCURY LNA SYBR Green PCR Kit (200) (Cat No: 339345) PAXgene Blood miRNA Kit (50) (Cat No: 763134) miRNeasy Serum/Plasma Kit (50) (Cat No: 217184) PCR Tubes 0.2 ml (1000) (Cat No: 981005) TF/10UL FILTER TIPS FOR P-10,RAC (Cat No: TF-10-R-S) TF/100UL FILTER TIPS FOR (Cat No: TF-100-R-S) TF /1000UL UNIVERSAL FILTER TIPS (Cat No: TF-1000-R-S)

Kit and consumables required for DNA methylation analysis:

ZymoResearch EZ DNA Methylation-Gold™ Kit 200 Preps (Cat no: D5006) ZymoResearch Human Methylated & Non-methylated DNA Set (DNA w/ primers) 1 set (Cat no: D5014) ZymoResearch ZymoTaq qPCR Premix 200 Reactions (Cat no: E2055) Primary synthesis consumable for 1 gene region AXYGEN 0.5ml Thin Wall PCR Tubes,Flat Cap. Clear1000 (Cat no: PCR-05-C) Capp 2.0ml Boil-Proof Microtubes. Clear 1000 (Cat no: MCT-200-C) Capp 10 ul Dnase, Rnase Free Bulk Pipet tips 10 rack (Cat no: 5.030.010) Capp 200 ul Dnase, Rnase Free Bulk Pipet ucu (Yellow Tips) 10 rack (Cat no: 4.130.075) Capp 1000 ul Dnase, Rnase Free Bulk Pipet ucu (Blue Tips) 10 rack (Cat no: 4.130.135) Bio Molecular Systems Mic Tubes and Caps 1 Box: 20 racks of 48 tubes/rack, 960 Tubes in Strips of 4 with matching caps (Cat no: MIC-TUBES960).

The motivation element behind the choice of miRNAs in the current work is a product of the following integrated online databases for miRNA target prediction and functional analysis.http://microrna.osumc.edu, https://www.genecards.org. http://www.mirdb.org/miRDB/ Gene association networks with ACE2, TMPRSS2, PARP, HOX1 genes in COVID 19 cases were analyzed using GeneMANIA (Multiple Association Network Integration Algorithm) for prediction of possible functional interactions among them (http://www. genemania.org).

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 18 and 65 included will suffer from COVID 19, and specific treatment should not yet be initiated.
* COVID 19 diagnosis of patients will be based on full medical history, thorough clinical examination, radiological imaging, laboratory assessment, and SARS-CoV-2 analysis by RT-PCR.

Exclusion Criteria:

* People with chronic lung disease or previous AC surgery
* People with immune deficiency or cancer patients
* Patients receiving immunosuppressive therapy for autoimmune disease
* People with neurological diseases affecting the respiratory muscles, such as hypotonia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: On the basis of the inclusion and exclusion criteria 105 patients subjects will be included in this study, divided into three groups; group I (n = 35) patients are mild, group II (n = 35) patients are moderate, and group III (n = 35) patients are severe and critical. Mild and moderate cases are usually defined as those without severe pneumonia or sever acute respiratory syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the relationship between the severity of disease and epigenetic factors in COVID 19 | Seven months
  Analysis of pathway-related micro RNAs in patients with mild, moderate and severe Covid 19 clinics

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan T. Adas, Prof, Study Director — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Asuman Gedikbasi, Assoc.Prof., Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Kadriye Yaşar, Prof., Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Nilgün Isiksacan, Assoc.Prof., Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Zafer Çukurova, Assoc.Prof., Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Oya G. Hergünsel, MD, Intensivist, Principal Investigator — Bakirkoy Dr. Sadi Konuk Research and Training Hospital; Sacide Pehlivan, Prof., Principal Investigator — Istanbul University
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Since studies on COVID 19 in our country during this pandemic are subject to certain permissions, the decision will be made when the permit processes are completed.